CLINICAL TRIAL: NCT02571673
Title: Feasibility Study of the Head and Neck Survivorship Tool: Assessment and Recommendations (HN-STAR)
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Columbia University (Other); Hartford Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 15-245
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Cancer
Keywords: Survivorship; Quality of Life; HN-STAR web-based; 15-245
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Survivors of head and neck cancer: Data collection will take place in two parts. Aim 1: Part 1 will enroll 10 patients at MSK to participate in component pilot testing and usability testing of HN-STAR and the associated surveys. We will also elicit feedback from the NP. After incorporating any changes to HN-STAR or the surveys based on findings from Aim 1: Part 1, Aim 1: Part 2 will enroll 30 additional patients from MSK and 15 from HH to provide feedback on usability. We will also survey each patient's PCP in Aim 1: Part 2.
  Interventions: Behavioral: Assessments

INTERVENTIONS:
Behavioral: Assessments — Usability outcomes will come from patient surveys and interviews and a nurse practitioner interview in Aim 1: Part 1. In Aim 1: Part 2, patients and their primary care providers will complete online surveys regarding feasibility. Health outcomes and data regarding health care actions will be collected from HN-STAR and the clinic note will be collected to assess feasibility of collecting these metrics in a future trial. Directly after each clinic visit, the NP will complete one brief online survey for each participant.

SUMMARY:
This study is being done to understand how survivors of head and neck cancer think they can make HN-STAR (the Survivor Self-Assessment, the survivorship clinic experience, and the Survivorship Care Plan the best it can be. Once the investigators have your input and input from other survivors, they can make changes to HN-STAR, so that they can test this tool in a larger study. The larger study will tell them whether using HN-STAR improves the care of head and neck cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

Aim 1: Part 1

* Have completed treatment for head and neck cancer at least 1 year prior to survivorship visit and have no evidence of disease
* Have a primary care provider
* Be able to provide informed consent
* Be able to speak and read English
* Be at least 18 years old

Aim 1: Part 2

* Have completed treatment for head and neck cancer at least 1 year prior to survivorship visit and have no evidence of disease
* Have a primary care provider
* Be able to provide informed consent
* Be able to speak and read English
* Be at least 18 years old

Exclusion Criteria:

Aim 1: Parts 1 and 2 is the same

* Patients or providers who cannot speak or read English
* Patients with cognitive, visual, or motor impairment such that they cannot complete the Survivor Self-Assessment as assessed by the research team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinics
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Talya Salz, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Salz T, McCabe MS, Oeffinger KC, Corcoran S, Vickers AJ, Salner AL, Dornelas E, Schnall R, Raghunathan NJ, Fortier E, Baxi SS. A head and neck cancer intervention for use in survivorship clinics: a protocol for a feasibility study. Pilot Feasibility Stud. 2016 May 5;2:23. doi: 10.1186/s40814-016-0061-3. eCollection 2016. PMID 27965842
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Survivors of Head and Neck Cancer: Participants must have completed treatment for head and neck cancer at least 1 year prior to survivorship visit and have no evidence of disease.
Period: Overall Study
Arm/Group | Survivors of Head and Neck Cancer
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Survivors of Head and Neck Cancer
Number analyzed (Participants) | 65
Age, Continuous [Median (Full Range); unit: years] | 60 [29 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 65
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 57
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Recommendations for Cancer Surveillance (Patient-reported Outcomes From the Survivor Self-Assessment)
Description: Using data from survivors in Aim 1: Part 2 (N=45), we will abstract data on health care actions from both the medical record and HN-STAR. Such data include receipt of appropriate oncologic surveillance, identification and management of symptoms, and appropriate preventive health services, as indicated by referrals, prescriptions, and recommendations in both clinic notes and the HN-STAR Survivor Self-Assessment. For each participant, HN-STAR generates a Treatment Summary/TS for the clinician to review and verify its accuracy compared with clinical documentation with the participant medical record.
Time Frame: 2 years
Measure: Number; unit: % of pts w/accurate TS for primary site
Arm/Group | Survivors of Head and Neck Cancer
Number analyzed (Participants) | 45
% of pts w/accurate TS for primary site | 93

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Survivors of Head and Neck Cancer
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT02571673/Prot_SAP_001.pdf
  • Informed Consent Form (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT02571673/ICF_000.pdf